CLINICAL TRIAL: NCT06834230
Title: Effect of Dotinurad in Hyperuricemia With Hypertension: a Randomized Study With Febuxostat (DIANA-NEXT)
Brief Title: Effect of Dotinurad in Hyperuricemia With Hypertension
Acronym: DIANA-NEXT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Saga University (Other)
Responsible Party: Principal Investigator, Koichi Node, Professor, Saga University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00003
Record Dates: First submitted 2025-01-30; First posted 2025-02-19 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Hyperuricemia or Gout; Hypertension
Keywords: Febuxostat; Dotinurad; CAVI; Arterial stiffness
MeSH Terms: conditions — Hyperuricemia; Gout; Hypertension | interventions — dotinurad; Febuxostat

STUDY DESIGN:
Intervention Model Description: Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dotinurad (Experimental): Start at 0.5 mg once daily, and then referring to the attached document and the following dosage examples, gradually increase the dose to the maintenance dose (2 mg once daily).
  Interventions: Drug: Dotinurad
- Febuxostat (Active Comparator): Start at 10 mg once daily, and then referring to the attached document and the following dosage examples, gradually increase the dose to the maintenance dose (40 mg once daily).
  Interventions: Drug: Febuxostat

INTERVENTIONS:
Drug: Dotinurad — Start at 0.5 mg once daily, and then referring to the attached document, gradually increase the dose to the maintenance dose (2 mg once daily).
  Other Names: URECE
  Arms: Dotinurad
Drug: Febuxostat — Start at 10 mg once daily, and then referring to the attached document, gradually increase the dose to the maintenance dose (40 mg once daily).
  Other Names: Feburic
  Arms: Febuxostat

SUMMARY:
The effect of dotinurad on CAVI (cardio-ankle vascular index) will be compared with that of febuxostat in patients with hyperuricemia complicated by hypertension.

DETAILED DESCRIPTION:
After determining eligibility of patients for whom consent is obtained, all patients who meet the eligibility criteria will be enrolled and randomized to one of two groups: dotinurad or febuxostat. In principle, a baseline (0-week) examination will be conducted within 70days after obtaining consent, followed by 24 weeks of observation and examination. During the observation period, no changes or additions to the dosage or administration of drugs other than the study drug will be made in principle, but changes or additions will be permitted under the overall clinical judgment of the physician in charge according to the medical conditions of the study participants.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 20 years or older at the time of consent (regardless of gender)
2. Patients with hyperuricemia with serum uric acid level >7.0 mg/dL who have not received any urate lowering drug within 27 days prior to obtaining consent, or patients who were receiving urate lowering drugs at the time of obtaining consent but have been off the drugs for more than 27 days
3. Hypertensive patients who meet the definition of hypertension in the latest Hypertension Treatment Guidelines of the Japanese Society of Hypertension and whose treatment for hypertension (with or without drug therapy) has not changed within 4 weeks prior to eligibility determination
4. Patients who have given written consent to participate in this study

Exclusion Criteria:

1. Patients with unsettled gout after acute gouty arthritis
2. Patients currently suffering from urinary tract stones
3. Patients with known secondary hyperuricemia who have Lesch-Nyhan syndrome, hyperphosphoribosyl pyrophosphate synthase, congenital myogenic hyperuricemia, hematopoietic tumors (acute leukemia, malignant lymphoma, myeloproliferative disorders, myelodysplastic syndrome), solid tumors (breast cancer, seminoma, sarcoma, Wilms' tumor, small cell lung cancer), non-neoplastic diseases (psoriasis vulgaris, secondary polycythemia vera, hemolytic anemia), tumor melting syndrome, rhabdomyolysis, hypothyroidism, polycystic kidney disease, lead poisoning/lead nephropathy, Down syndrome, familial juvenile gout nephropathy, hyperlactatemia, or type 1 glycogenic disease
4. Patients with hypertensive emergencies and urgency
5. Patients with active malignancies
6. Patients with severe hepatic dysfunction
7. Patients with severe renal dysfunction with oliguria or anuria
8. Pregnant, possibly pregnant, or lactating patients
9. Patients with a history of hypersensitivity to the components of dotinurad and febuxostat
10. Patients receiving mercaptopurine hydrate or azathioprine
11. Other patients deemed inappropriate for this study by the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in CAVI | 24 weeks
  Change in CAVI at 24 weeks after study drug administration

SECONDARY OUTCOMES:
Change in CAVI category | 24 weeks
  Change in CAVI category (<8.0: normal, 8.0 to 9.0: borderline, 9.0 or greater: abnormal) at 24 weeks after study drug administration (key secondary endpoint)
Change in CAVI | 12 weeks
  Change in CAVI at 12 weeks after study drug administration
Change in CAVI category | 12 weeks
  Change in CAVI category (<8.0: normal, 8.0 to 9.0: borderline, 9.0 or greater: abnormal) at 12 weeks after study drug administration

OTHER OUTCOMES:
Changes in serum uric acid levels | 4, 8, 12 and 24 weeks
  Changes in serum uric acid levels at 4, 8, 12 and 24 weeks after study drug administration
Percentage of patients whose serum uric acid levels reach 6.0 mg/dL or less | 4, 8, 12 and 24 weeks
  Percentage of patients whose serum uric acid levels reach 6.0 mg/dL or less at 4, 8, 12, and 24 weeks after study drug administration
Change in AI | 24 weeks
  Change in AI at 24 weeks after study drug administration
Change in %MAP | 24 weeks
  Change in %MAP at 24 weeks after study drug administration
Change in serum NT-proBNP | 24 weeks
  Change in serum NT-proBNP at 24 weeks after study drug administration
Change in serum CRP | 24 weeks
  Change in serum CRP at 24 weeks after study drug administration
Change in serum oxidized LDL | 24 weeks
  Change in serum oxidized LDL at 24 weeks after study drug administration
Change in urinary albumin-creatinine ratio | 24 weeks
  Change in urinary albumin-creatinine ratio at 24 weeks after study drug administration
Change in urinary 8-OHdG | 24 weeks
  Change in urinary 8-OHdG at 24 weeks after study drug administration
Change in urinary NAG | 24 weeks
  Change in urinary NAG at 24 weeks after study drug administration
Changes in systolic and diastolic blood pressures | 12 and 24 weeks
  Changes in systolic and diastolic blood pressures at 12 and 24 weeks after study drug administration
Changes in pulse pressure (systolic blood pressure minus diastolic blood pressure) | 12 and 24 weeks
  Changes in pulse pressure (systolic blood pressure minus diastolic blood pressure) at 12 and 24 weeks after study drug administration
Changes in AST | 12 and 24 weeks
  Changes in AST at 12 and 24 weeks after study drug administration
Changes in ALT | 12 and 24 weeks
  Changes in ALT at 12 and 24 weeks after study drug administration
Changes inγ-GTP | 12 and 24 weeks
  Changes inγ-GTP at 12 and 24 weeks after study drug administration
Changes in HDL-C | 12 and 24 weeks
  Changes in HDL-C at 12 and 24 weeks after study drug administration
Changes in LDL-C | 12 and 24 weeks
  Changes in LDL-C at 12 and 24 weeks after study drug administration
Changes in TG | 12 and 24 weeks
  Changes in TG at 12 and 24 weeks after study drug administration
Changes in WBC (including fractions) | 12 and 24 weeks
  Changes in WBC (including fractions) at 12 and 24 weeks after study drug administration
Changes in PLT | 12 and 24 weeks
  Changes in PLT at 12 and 24 weeks after study drug administration
Changes in Cr | 12 and 24 weeks
  Changes in Cr at 12 and 24 weeks after study drug administration
Changes in eGFR | 12 and 24 weeks
  Changes in eGFR at 12 and 24 weeks after study drug administration
Changes in FIB-4 index | 12 and 24 weeks
  Changes FIB-4 index at 12 and 24 weeks after study drug administration
Change in echocardiographic parameters (LVEDV) | 24 weeks
  Change in LVEDV at 24 weeks after study drug administration
Changes in echocardiographic parameters (LVESV) | 24 weeks
  Changes in LVESV at 24 weeks after study drug administration
Change in echocardiographic parameters (LVEF) | 24 weeks
  Change in LVEF at 24 weeks after study drug administration
Change in echocardiographic parameters (septal e') | 24 weeks
  Change in septal e' at 24 weeks after study drug administration
Change in echocardiographic parameters (lateral e') | 24 weeks
  Change in lateral e' at 24 weeks after study drug administration
Change in echocardiographic parameters (mitral annular velocity (E)) | 24 weeks
  Change in mitral annular velocity (E) at 24 weeks after study drug administration
Change in echocardiographic parameters (E/e') | 24 weeks
  Change in E/e' at 24 weeks after study drug administration
Change in echocardiographic parameters (LVMI) | 24 weeks
  Change in LVMI at 24 weeks after study drug administration
Change in echocardiographic parameters (LAVI) | 24 weeks
  Change in LAVI at 24 weeks after study drug administration
Changes in protein levels as determined by proteomics analysis | 24 weeks
  Changes in protein levels as determined by proteomics analysis(Olink Target 96 Inflammation analysis, Olink Target 96 CVDⅡ analysis, Olink Target 96 CVDⅢ analysis) at 24 weeks after study drug administration
Adverse events | 24 weeks
  Adverse events that occurred after study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Koichi Node, Pr.,Dr., Principal Investigator — Saga University
Locations (1):
- Saga University, Saga, Saga-ken, Japan

IPD SHARING:
Plan to Share IPD: Undecided